CLINICAL TRIAL: NCT05576779
Title: Characterization of Early Patients Initiating Ofatumumab for Treatment of Multiple Sclerosis in the Real-World
Brief Title: Characterization of Early Patients Initiating Ofatumumab for Treatment of Multiple Sclerosis.
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: COMB157GUS11
Record Dates: First submitted 2022-10-10; First posted 2022-10-13 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Multiple Sclerosis
Keywords: Multiple sclerosis,; ofatumumab,; disease-modifying therapy,; COVID-19
MeSH Terms: conditions — Multiple Sclerosis; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- Ofatumumab: all eligible patients with at least 1 claim for ofatumumab observed during the index period were included in the ofatumumab cohort
  Interventions: Other: Ofatunumab
- Non-ofatumumab: patients with no evidence of ofatumumab during the index period were included in the non-ofatumumab cohort and included in subgroups based on the index medication: Siponimod, Ocrelizumab, Dimethyl fumarate, Glatiramer acetate

INTERVENTIONS:
Other: Ofatunumab — All eligible patients with at least 1 claim for ofatumumab observed during the index period were included in the ofatumumab cohort
  Groups: Ofatumumab

SUMMARY:
This was a retrospective cohort study utilizing secondary data from IQVIA's open source pharmacy claims database (i.e., IQVIA LRx) selecting patients with prescription claims for ofatumumab or other DMTs of interest.

DETAILED DESCRIPTION:
The date of first ofatumumab prescription claim or other DMT of interest was defined as the index date. No post-index requirements were imposed.

Patients were linked to IQVIA's open source medical claims databases (Dx) to obtain patient clinical characteristics.

The initial data were extracted in October 2020. The data and results were refreshed in April 2021 and July 2021 to allow for assessment of changes in characteristics at 6 and 9 months post-launch.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ≥ 1 prescription for ofatumumab in the LRx/Dx database were included. The date of the first observed prescription within the index window served as the index date.

  -. Patients with a diagnosis of COVID-19 or a COVID-19 vaccination any time during the study period.
* Patients with linkage to the Dx database.

Exclusion criteria

- No exclusion criteria were applied to patients in the study.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with prescription claims for ofatumumab or other DMTs of interest.
Sampling Method: Non-Probability Sample
Enrollment: 2101 (Actual)
Dates: Start 2020-12-03 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Proportion of patients initiating ofatumumab based on DMT use | 12-months prior to index date, where index date was defined as the date of first ofatumumab claim (or other DMT of interest for non-ofa cohorts)
  The primary measure was pre-index treatment status of patients initiating ofatumumab, measured as proportion (n, %) of DMT-naïve and DMT-experienced patients among patients initiating ofatumumab based on DMT use in the 12-month pre-index period.

SECONDARY OUTCOMES:
Age | Index date, defined as the date of first ofatumumab claim (or other DMT of interest for non-ofa cohorts)
  Age information was reported
Gender | Index date, defined as the date of first ofatumumab claim (or other DMT of interest for non-ofa cohorts)
  Gender information was reported
Number of patients: Geographic region | Index date, defined as the date of first ofatumumab claim (or other DMT of interest for non-ofa cohorts)
  Northeast, Midwest, South, West, Unknown
Number of patients: State level (Geographic region) | Index date, defined as the date of first ofatumumab claim (or other DMT of interest for non-ofa cohorts)
  The geographical heat map of ofatumumab utilization at the state level was presented.
Number of patients: Insurance type | Index date, defined as the date of first ofatumumab claim (or other DMT of interest for non-ofa cohorts)
  Cash, Commercial, Medicare, Medicare Part D, Medicaid, Unknown
Number of patients: Payer | Index date, defined as the date of first ofatumumab claim (or other DMT of interest for non-ofa cohorts)
  CVS, Aetna etc
Follow-up time | Variable Post-index period, where index date was defined as date of first ofatumumab claim (or other DMT of interest for non-ofa cohorts) (01/08/2019 - 31/05/2021)
  Ofatumumab persistence was assessed over the variable follow-up time.
Number of patients: Pre-index Charlson comorbidity index (CCI) | 12-months prior to index date, where index date was defined as the date of first ofatumumab claim (or other DMT of interest for non-ofa cohorts)
  Charlson Comorbidity Index predicts the ten-year mortality for a patient who may have a range of comorbid conditions. omorbidity was assessed using the Charlson Comorbidity Index (CCI), categorized as low (0-1) and high (≥2)
Number of patients: Pre-index comorbidities | 12-months prior to index date, where index date was defined as the date of first ofatumumab claim (or other DMT of interest for non-ofa cohorts)
  Number of patients with list of comorbidities were reported
Number of patients with a relapse in inpatient settings | 12-months prior to index date, where index date was defined as the date of first ofatumumab claim (or other DMT of interest for non-ofa cohorts)
  Number of patients with MS relapses were reported
Number of patients with a relapse in outpatient settings | 12-months prior to index date, where index date was defined as the date of first ofatumumab claim (or other DMT of interest for non-ofa cohorts)
  Number of patients with MS relapses were reported
Number of relapses in all patients | 12-months prior to index date, where index date was defined as the date of first ofatumumab claim (or other DMT of interest for non-ofa cohorts)
  Number of patients with MS relapses were reported
Number of relapses in patients with at least 1 relapse | 12-months prior to index date, where index date was defined as the date of first ofatumumab claim (or other DMT of interest for non-ofa cohorts)
  Number of patients with MS relapses were reported
Claims-Based Disability Score | 12-months prior to index date, where index date was defined as the date of first ofatumumab claim (or other DMT of interest for non-ofa cohorts)
  Pre-index MS-related symptoms and secondary conditions (n, %) based on a Claims-Based Disability Score (e.g., sensory problems, eye symptoms, pyramidal symptoms, bladder/bowel symptoms, fatigue/malaise, muscular weakness, durable medical equipment utilization.
Number of pre-index Brain and Spinal MRI scans | 12-months prior to index date, where index date was defined as the date of first ofatumumab claim (or other DMT of interest for non-ofa cohorts)
  Categorized as: No MRI, 1, 2, 3+
Number of patients: Hepatitis B virus screening | 12-months prior to index date, where index date was defined as the date of first ofatumumab claim (or other DMT of interest for non-ofa cohorts)
  Yes/No
Number of patients: Quantitative serum immunoglobulin screening | 12-months prior to index date, where index date was defined as the date of first ofatumumab claim (or other DMT of interest for non-ofa cohorts)
  Yes/No
Number of patients: Pre-index flu shot | 12-months prior to index date, where index date was defined as the date of first ofatumumab claim (or other DMT of interest for non-ofa cohorts)
  Yes/No
Number of patients: Post-index flu shot | Variable Post-index period, where index date was defined as Date of first ofatumumab claim (or other DMT of interest for non-ofa cohorts) (01/08/2019 - 31/05/2021)
  Yes/No
Pre-index: Number of patients with COVID-19 diagnosis | 12-months prior to index date, where index date was defined as the date of first ofatumumab claim (or other DMT of interest for non-ofa cohorts)
  Yes/No
Post-index: Number of patients with COVID-19 diagnosis | Variable Post-index period, where index date was defined as Date of first ofatumumab claim (or other DMT of interest for non-ofa cohorts) (01/08/2019 - 31/05/2021)
  Yes/No
Days between COVID-19 diagnosis and initiation of ofatumumab | Variable Post-index period, where index date was defined as Date of first ofatumumab claim (or other DMT of interest for non-ofa cohorts) (01/08/2019 - 31/05/2021)
  Days between COVID-19 diagnosis and initiation of ofatumumab were reported
Pre-index: Number of patients with COVID-19 vaccination | 12-months prior to index date, where index date was defined as the date of first ofatumumab claim (or other DMT of interest for non-ofa cohorts)
  Yes/No
Post-index: Number of patients with COVID-19 vaccination | Variable Post-index period, where index date was defined as Date of first ofatumumab claim (or other DMT of interest for non-ofa cohorts) (01/08/2019 - 31/05/2021)
  Yes/No
Days between COVID-19 vaccination and initiation of ofatumumab | Variable Post-index period, where index date was defined as Date of first ofatumumab claim (or other DMT of interest for non-ofa cohorts) (01/08/2019 - 31/05/2021)
  Days between COVID-19 vaccination and initiation of ofatumumab were reported.
Proportion of patients with steroid use or antihistamine as pre-medication with ofatumumab first dose | Variable Post-index period, where index date was defined as Date of first ofatumumab claim (or other DMT of interest for non-ofa cohorts) (01/08/2019 - 31/05/2021)
  E.g. diphenhydramine, dexamethasone and other steroids. pre-medication was defined as medication observed within two days of ofatumumab initiation.
Pre-index HCRU: Number of patients with an inpatient visit | 12-months prior to index date, where index date was defined as the date of first ofatumumab claim (or other DMT of interest for non-ofa cohorts)
  Number of patients with an inpatient visits were reported to report the pre-index healthcare resource utilization
Pre-index HCRU: Number of patients with an ED visit | 12-months prior to index date, where index date was defined as the date of first ofatumumab claim (or other DMT of interest for non-ofa cohorts)
  Number of patients with an ED visit were reported to report the pre-index healthcare resource utilization
Pre-index HCRU: Number of patients with an outpatient visit | 12-months prior to index date, where index date was defined as the date of first ofatumumab claim (or other DMT of interest for non-ofa cohorts)
  Number of patients with an outpatient visit were reported to report the pre-index healthcare resource utilization
Pre-index HCRU: Number of patients with a pharmacy claim | 12-months prior to index date, where index date was defined as the date of first ofatumumab claim (or other DMT of interest for non-ofa cohorts)
  Number of patients with a pharmacy claim were reported to report the pre-index healthcare resource utilization
Post-index HCRU: Number of patients with an inpatient visit | Variable Post-index period, where index date was defined as Date of first ofatumumab claim (or other DMT of interest for non-ofa cohorts) (01/08/2019 - 31/05/2021)
  Number of patients with an inpatient visits were reported to report the post-index healthcare resource utilization accrued while on ofatumumab
Post-index HCRU: Number of patients with an ED visit | Variable Post-index period, where index date was defined as Date of first ofatumumab claim (or other DMT of interest for non-ofa cohorts) (01/08/2019 - 31/05/2021)
  Number of patients with an ED visit were reported to report the post-index healthcare resource utilization accrued while on ofatumumab
Post-index HCRU: Number of patients with an outpatient visit | Variable Post-index period, where index date was defined as Date of first ofatumumab claim (or other DMT of interest for non-ofa cohorts) (01/08/2019 - 31/05/2021)
  Number of patients with an outpatient visit were reported to report the post-index healthcare resource utilization accrued while on ofatumumab
Post-index HCRU: Number of patients with a pharmacy claim | Variable Post-index period, where index date was defined as Date of first ofatumumab claim (or other DMT of interest for non-ofa cohorts) (01/08/2019 - 31/05/2021)
  Number of patients with a pharmacy claim were reported to report the post-index healthcare resource utilization accrued while on ofatumumab

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, East Hanover, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Results for COMB157GUS11 from the Novartis Clinical Trials Website — http://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=17981